CLINICAL TRIAL: NCT06996873
Title: Management Of Aggressive Spinal Hemangioma
Brief Title: Aggressive Spinal Hemangioma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Momen Ahmed Mohamed Kamel, resident at the Orthopaedic and Trauma Surgery department, Assiut University
Other Study IDs: Spinal Hemangioma mangement
Record Dates: First submitted 2025-04-02; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Aggressive Spinal Hemangiomas
Keywords: hemangiomas; management
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with symptomatic, radiologically confirmed aggressive spinal hemangiomas treated at Assiut: Confirmed diagnosis of aggressive vertebral hemangioma via imaging (MRI/MSCT) and clinical symptoms (e.g., pain, neurological deficits).

SUMMARY:
This research is a case series analysis to evaluate aggressive vertebral hemangiomas. It focuses on clinical presentation, diagnostic imaging accuracy (X-ray, MRI, MSCT, angiography), and treatment efficacy. The primary goal is to establish optimal management protocols.

DETAILED DESCRIPTION:
Hybrid methodology integrating retrospective case reviews (from Assiut University Hospital's Orthopedic Surgery Department) with synthesis of existing literature.

Objectives:

Characterize clinical presentations and imaging findings. Compare diagnostic accuracy across modalities. Analyze treatment outcomes, including procedural success rates and complications.

Tools:

Imaging: X-ray for initial screening, MRI/MSCT for soft tissue and spinal cord involvement, angiography for vascular mapping.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with aggressive spinal hemangiomas based on clinical symptoms and imaging findings.
* Cases confirmed through diagnostic modalities such as X-ray, MRI, MSCT, or angiography.
* Patients presenting with symptoms such as pain, neurological deficits, or spinal instability attributable to the hemangioma.

Exclusion Criteria:

* Patients with incidentally discovered spinal hemangiomas (asymptomatic cases found during evaluations for unrelated conditions).
* Cases lacking sufficient diagnostic evidence to confirm aggressive spinal hemangioma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic, radiologically confirmed aggressive spinal hemangiomas treated at Assiut University Hospital. Excludes incidentally discovered cases.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Neurological Symptom Resolution | 3 months
  using the Pain intensity (VAS scale)

SECONDARY OUTCOMES:
Functional Status Improvement | 3 months
  using ASIA Impairment Scale (primary)
  Threshold: ≥1-grade improvement on ASIA scale sustained for ≥3 months